CLINICAL TRIAL: NCT05842551
Title: The Effect of Prismatic Lenses in Association With tDCS in Patients With Neglect: a Pilot Study
Brief Title: Prismatic Lenses and tDCS in Neglect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda USL Toscana Sud Est (Other Government)
Responsible Party: Principal Investigator, Simona Spaccavento, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1183
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Ischemic
Keywords: stroke; neglect; tDCS; prismatic lenses
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Patients will receive anodic tEs combined with prismatic lenses for two weeks
  Interventions: Combination Product: Prismatic adaptation and electric stimulation
- Control (Sham Comparator): Patients will receive sham tEs combined with prismatic lenses for two weeks
  Interventions: Combination Product: Prismatic adaptation and electric stimulation

INTERVENTIONS:
Combination Product: Prismatic adaptation and electric stimulation — Combinatory effect of tEs and prismatic lenses in the experimental group and of sham stimulation and prismatic lenses in control group

SUMMARY:
The goal of this study is to to evaluate the effect and feasibility of a rehabilitation protocol with prismatic lenses associated with tDCS, compared to a prismatic lens rehabilitation protocol associated with sham stimulation, in reducing the signs of neglect in a group of patients with spatial heminegligence following ischemic stroke of the right hemisphere.

The secondary objective is to evaluate the impact of this rehabilitation protocol on functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* ischemic stroke
* hospitalization within 90 days of the event

Exclusion Criteria:

* heamorrhagic stroke
* history of neurological disease
* history of psychiatric disease
* use of alchool and drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological outcome | Change from baseline OCS at 2 weeks
  Oxford Cognitive Screening (OCS): is structured in 10 subtests: picture naming (0-4); semantics (0-3); orientation (0-4); visual field (0-4); sentence reading (0-15); number writing (0-3); calculation (0-4); broken hearts (0-50); praxis (0-12); recall and recognition (0-4); trails task (0-13)
Neuropsychological outcome | Change form baseline the semi structured scale for the functional evaluation of extrapersonal neglect at 2 weeks
  The semi structured scale for the functional evaluation of extrapersonal neglect (0-9); high score means a worse outcome
Neuropsychological outcome | Change form baseline the semi structured scale for the functional evaluation of personal neglect at 2 weeks
  The semi structured scale for the functional evaluation of personal neglect (0-9); high score means worse outcome
Neuropsychological outcome | Change from baseline the Bergegò Scale at 2 weeks.
  Bergegò Scale (0-30); high score means a better outcome
Functional outcome | Change from baseline the Barthel Index at 2 weeks
  Barthel Index (0-100); high score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simona Spaccavento, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri, Bari, Ba, Italy